CLINICAL TRIAL: NCT00265694
Title: A Randomized Phase III Trial of Vinorelbine Versus Gemcitabine and Carboplatin for Elderly Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Random Trial for Elderly Patients With NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INJE05-06
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2005-12-15 (Estimated); Status verified 2005-06

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine; Gemcitabine; Carboplatin

INTERVENTIONS:
Drug: vinorelbine, gemcitabine and carboplatin

SUMMARY:
1. Recently a radomized trial of vinorelbine versus best supportive care in patients at 70 years of age or older demonstrated a definite improvement in overall survival rate and quality of life with chemotherapy.
2. The role of combination therapy containing the platinum compound, which is the standard therapy for the young patients is still vague.
3. Gemcitabine and carboplatin have favorable toxicity profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed, advanced(clinical stage IIIB or IV) NSCLC
* No previous chemotherapy history
* Age ≥ 65 years
* ECOG performance status ≤ 2
* Adequate marrow function (ANC ≥ 2,000/mm3, platelet ≥ 100,000/mm3), renal and liver function (total bilirubin < 2.0 mg/dL, AST/ALT levels < 3 × the upper limit of normal, serum creatinine < 2.0 mg/dL)
* Patients with informed written consent

Exclusion Criteria:

* Patients with other major illness(active infection, severe heart disease, concomitant malignancy, etc)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Young Jin Yuh, M.D., Principal Investigator
Locations (1):
- Inje University Sanggyepaik Hospital, Seoul, South Korea